CLINICAL TRIAL: NCT04838977
Title: Pediatric Injury: Modules to Manage Medical Stress
Brief Title: Recovery After Stress Toolkit (RESET) Study
Acronym: ReSeT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HD096350; R24HD096350 (NIH)
Record Dates: First submitted 2021-03-30; First posted 2021-04-09 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Post-Traumatic Stress Disorder in Children; Post-Traumatic Stress Disorder in Adolescence

STUDY DESIGN:
Intervention Model Description: Study comparing treatment to usual care.
Who Masked: Investigator
Masking Description: Investigators will not be aware of study assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RESET (Experimental): Children will view 8 educational modules online and participate in 8 sessions with a therapist via telehealth.
  Interventions: Behavioral: RESET
- Control (No Intervention): Children will receive usual post-trauma care.

INTERVENTIONS:
Behavioral: RESET — Therapy
  Arms: RESET

SUMMARY:
This study evaluates the use of web-based educational modules combined with telehealth delivered therapy for children with post-traumatic stress symptoms (PTSS) after receiving hospital based medical attention for an injury. Half of the participants will received the online therapy and half of the participants will receive usual care.

DETAILED DESCRIPTION:
As many as 30% of children develop post-traumatic stress symptoms after an injury. Post-traumatic stress symptoms can decrease children's quality of life. Psychological distress may emerge after the child is discharged from the hospital and may go unrecognized. Cognitive behavioral therapy and graduated exposures are standard treatments for PTSS.

ELIGIBILITY:
Inclusion Criteria:

* 8 years to 17 years at enrollment
* Treated for an injury in the ED or hospitalized
* Abbreviated Injury Scale (AIS) score 2 or greater
* Parent and child English speaking
* Broad band internet availability at home
* Residing with parent or legal guardian

Exclusion Criteria:

* Moderate or severe traumatic brain injury (GCS less than 13)
* Diagnosed with moderate or severe intellectual disability
* Pre-existing psychiatric disorder that required hospitalization
* Abuse or interpersonal injury as mechanism of injury
* Currently receiving psychotherapy
* Hospitalized for injury over 30 ays
* Death of a family member or friend at time of injury

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather T Keenan, MDCM, Principal Investigator — University of Utah
Locations (3):
- United States (3):
  - Cincinnati CHildren's Hospital, Cincinnati, Ohio
  - University of Texas Health Sciences Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified participant data underlying the trial will be made available 3 years after the last enrolled subject has completed all procedures to investigators who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP
Time Frame: 36 months after last subject has completed all procedures. Data will be available for 36 months.
Access Criteria: Investigators who provide a methodologically sound proposal

REFERENCES:
- [Derived] Keenan HT, Wade SL, Miron D, Presson AP, Clark AE, Ewing-Cobbs L. Reducing Stress after Trauma (ReSeT): study protocol for a randomized, controlled trial of an online psychoeducational program and video therapy sessions for children hospitalized after trauma. Trials. 2023 Nov 28;24(1):766. doi: 10.1186/s13063-023-07806-y. PMID 38017574

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 93 children randomized
Pre-assignment Details: 130 children eligible for randomization No consent obtained = 37
  Reasons:
  Currently receiving psychotherapy (exclusion criteria), n=5 Parent felt too much time required, n=6 Participant no longer interested, n=9 No reason given/unknown, n=8 Other reason, n=9
Period: Overall Study
Arm/Group | RESET | Control
Started | 47 | 46
Completed | 44 | 42
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RESET | Control | Total
Number analyzed (Participants) | 47 | 46 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 47 | 46 | 93
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.6 (2.4) | 11.7 (2.5) | 11.65 (2.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 22 | 37
  Male | 32 | 24 | 56
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 46 | 93
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 35 | 37 | 72
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 17 | 26
  Not Hispanic or Latino | 37 | 29 | 66
  Unknown or Not Reported | 1 | 0 | 1
CPSS [Mean (Standard Deviation); unit: CPSS score] — We measured the combined parent-child CPSS prior to randomization which served as the baseline.
  CPSS score | 22.7 (9.4) | 23.7 (8.6) | 23.2 (9.0)

OUTCOME MEASURES:

1. Primary Outcome: Child PTSD Symptom Scale (CPSS)
Description: 17 items listing potential PTSD symptoms scored on a Likert scale of 0 to 3 with 0=Not at all and 3= 5 or more times a week. 7 additional yes/no questions ask if problems interfered with various activities. Higher score is worse. Range 0 to 80. We used the combined child report and parent report. The highest item score from either parent or child was summed.
Time Frame: 10 weeks post-randomization
Population: We had 3 children not complete the intervention and 4 controls not complete the final data collection as shown in participant flow.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RESET | Control
Number analyzed (Participants) | 44 | 42
Score on a scale | 10.4 (8.5) | 14 (9.5)
Statistical Analysis 1: Comparison: RESET vs Control; The null hypothesis is there is no difference in mean CPSS at 10 weeks in the intervention group versus the control group; Test type: Superiority; Between group difference = -4.2, 95% CI 2-sided [-7.6 to -0.8]

2. Secondary Outcome: Screen for Anxiety Related Emotional Disorders (SCARED)
Description: 41-item survey with three point Likert scale responses (not sure, somewhat true, very true) that asks about common difficulties for children with anxiety. Higher scores indicate worse outcomes. Range 0-82
Time Frame: 10 weeks post-randomization
Population: Some participants did not complete the measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RESET | Control
Number analyzed (Participants) | 38 | 33
Score on a scale | 12.6 (12.4) | 20.8 (14.7)

3. Secondary Outcome: Patient Reported Outcome Measurement Information System (PROMIS) Pediatric Depressive Symptoms
Description: PROMIS pediatric item bank : 8 questions with a 5-point Likert response from Never to Almost Always. Higher scores means more depressive symptoms. T-score with mean = 50; Standard Deviation (SD)=10.
Time Frame: 10-weeks post-randomization
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RESET | Control
Number analyzed (Participants) | 42 | 42
Score on a scale | 42.9 (9.0) | 49.8 (10.9)

4. Secondary Outcome: Pediatric Quality of Life Inventory (PedsQL)
Description: 15 question scale based on physical, emotional, social and school functioning answered on a 5-point Likert scale (never to almost always). Score is 0 - 100 with higher scores indicating better HRQoL. Parent proxy scale.
Time Frame: 10-weeks
Population: Some participants did not complete all scales.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RESET | Control
Number analyzed (Participants) | 43 | 40
Score on a scale | 71.4 (16.7) | 68.4 (17.2)

5. Other Pre Specified Outcome: Connor David Resilience Scale
Description: 10-item scale with LIkert response from 0 - not true to 4=true nearly all of the time. Range is 0 to 40 with higher scores indicating more resilience (better).
Time Frame: 10-weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RESET | Control
Number analyzed (Participants) | 40 | 41
Score on a scale | 26.8 (12.1) | 21.4 (10.5)

6. Other Pre Specified Outcome: PROMIS Pediatric Anger
Description: 5 question PROMIS measure answered with a 5-point Likert scale. A higher score indicates more anger (worse). T-score with mean = 50; SD = 10.
Time Frame: 10-weeks post-randomization
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RESET | Control
Number analyzed (Participants) | 42 | 42
Score on a scale | 43.6 (11.3) | 47.9 (11.9)

7. Other Pre Specified Outcome: PROMIS Pediatric Psychological Stress Experience
Description: 8-question PROMIS measure answered with a 5-point Likert scale. A higher score is more stress (worse). T-score with mean 50; SD 10.
Time Frame: 10-weeks post-randomization
Population: Not all children completed all measures.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RESET | Control
Number analyzed (Participants) | 42 | 42
Score on a scale | 47.1 (9.8) | 54.2 (10.8)

8. Other Pre Specified Outcome: PROMIS Pediatric Physical Stress Experience
Description: 8-question PROMIS measure answered on a 5-point Likert scale. A higher score is more physical stress (worse). T-score with mean 50; SD 10.
Time Frame: 10-weeks
Population: Not all children completed all of the measures.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RESET | Control
Number analyzed (Participants) | 42 | 42
Score on a scale | 47.4 (9.6) | 53.3 (9.7)

9. Other Pre Specified Outcome: PROMIS Pediatric Anxiety
Description: 8-question PROMIS measure answered on a 5-point LIkert scale. A higher score is more anxiety (worse). T-score with mean 50; SD 10.
Time Frame: 10-weeks
Population: Not all children completed all of the measures.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RESET | Control
Number analyzed (Participants) | 42 | 42
Score on a scale | 42.7 (11.2) | 47.5 (11.1)

10. Other Pre Specified Outcome: PROMIS Pediatric Global Health
Description: Seven questions about global health with 5-point Likert response from excellent to poor. A higher score is more poor health (worse). T-score with mean 50; SD 10.
Time Frame: 10-weeks
Population: Not all children completed all of the measures.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RESET | Control
Number analyzed (Participants) | 42 | 42
Score on a scale | 51.0 (9.9) | 47 (10.7)

ADVERSE EVENTS:
Time Frame: From enrollment in the trial until completion of therapy or at 10 weeks dependent on arm.
Groups:
- Control: Children will receive usual post-trauma care.
  Control: Usual care
Arm/Group | Control | RESET
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/47
Other Adverse Events (participants affected / at risk) | 0/46 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT04838977/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT04838977/ICF_000.pdf